CLINICAL TRIAL: NCT00910494
Title: Intraoperative Radiotherapy (IORT) for Rectal Cancer Using the Photon Radiosurgery System (PRS): A Phase I Clinical Trial
Brief Title: Intraoperative Radiotherapy for Rectal Cancer Using the Photon Radiosurgery System
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: No longer practical to deliver treatment
Sponsor: University of Dundee (Other)
Responsible Party: Principal Investigator, Ian Sanders, Specialist Registrar, University of Dundee
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EB/JK/LET/LN1277
Record Dates: First submitted 2009-05-28; First posted 2009-06-01 (Estimated); Last update posted 2018-04-24 (Actual); Status verified 2018-04

CONDITIONS: Rectal Neoplasm
Keywords: Rectal neoplasm C04.588.274.476.411.307.790; Intraoperative Radiotherapy
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 12 Gray IORT (Experimental)
  Interventions: Radiation: Photon Radiosurgery System IORT
- 15 Gray IORT (Experimental)
  Interventions: Radiation: Photon Radiosurgery System IORT

INTERVENTIONS:
Radiation: Photon Radiosurgery System IORT
  Arms: 12 Gray IORT
Radiation: Photon Radiosurgery System IORT
  Arms: 15 Gray IORT

SUMMARY:
The investigators would like to test the safety and efficacy of intraoperative radiotherapy (IORT) in rectal cancer using the Photon Radiosurgery System (PRS).

DETAILED DESCRIPTION:
Rectal cancer is usually managed by a combination of surgery and x-ray treatments (radiotherapy). The standard way of delivering radiotherapy is with external 'beams' directed at the tumour site. However, although in rectal cancer these treatments are effective, patients are often troubled by late side effects. An alternative option is to deliver the x-rays at the same time as surgery. This is known as intraoperative radiotherapy, or IORT, and a number of techniques have already been tried. There is a new IORT technology known as the Photon Radiosurgery System (PRS) which we are using to treat breast and brain cancers. Our experience to date has informed us that IORT with this x-ray source is safe and effective. We would like to use the technology to treat rectal cancer and believe that it may improve disease outcomes without the side effects associated with standard radiotherapy. We would also like to study the biological processes that follow radiation. It is not understood why some people are more sensitive to x-ray treatments than others. If we knew the reasons for this then we might be able to individualise treatments.

ELIGIBILITY:
Inclusion Criteria:

* Operable rectal cancer

Exclusion Criteria:

* Locally advanced disease requiring long course pre-operative chemoradiation, metastatic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2010-01; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
surgical complication rate | 30 days post treatment

SECONDARY OUTCOMES:
survival | 5 year
local control | 5 year

CONTACTS AND LOCATIONS:
Overall Officials: Alastair Munro, MBChB, Principal Investigator — University of Dundee
Locations (1):
- University of Dundee, Dundee, Tayside, United Kingdom